CLINICAL TRIAL: NCT00612599
Title: Comparison of the Pharmacodynamics and Pharmacokinetics of Biphasic Insulin Aspart 50 to Biphasic Insulin Aspart 70 in Non-obese and Obese With Type 2 Diabetes Mellitus
Brief Title: Comparison of Pharmacodynamics and Pharmacokinetics of Biphasic Insulin Aspart 50 to Biphasic Insulin Aspart 70 in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1526
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
  Other Names: BIASP

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the pharmacodynamics and pharmacokinetics of biphasic insulin aspart 50 three times a day to biphasic insulin aspart 70 three times a day in non-obese and obese with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months
* Stable glycaemic control, having been on the existing treatment for at least 1 month
* BMI between 23-28 kg/m2 (non-obese) or between 30-35 kg/m2 (obese)
* HbA1c below 9.0%
* Willing to eat three main meals per day during the trial period and perform Self-Monitoring of Blood Glucose (SBGM) regularly

Exclusion Criteria:

* A history of drug abuse or alcohol dependence
* Blood donation within the last 3 months
* Currently being treated with systemic corticosteroids, Mono Amine Oxidase (MAO) inhibitors, beta-adrenergic blocking agents, anabolic steroids or any other drug affecting blood glucose
* Severe, uncontrolled hypertension
* Proliferative retinopathy or maculopathy requiring acute treatment
* Pregnancy, breast-feeding, intention of becoming pregnant or judged not to be using adequate contraceptive measures (for women of childbearing potential only contraceptive pills and intra uterine devices are considered as adequate contraceptive methods)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-09; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Area under the serum glucose concentration profile during 24 hours | after 4 weeks of treatment

SECONDARY OUTCOMES:
Pharmacodynamics properties
Pharmacokinetic properties
8-point self-monitored blood glucose profiles
Adverse events
Hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Århus C, Denmark

REFERENCES:
- [Result] Parkner T, Dyrskog SE, Laursen T, Chen JW, Mouritzen U, Brondsted L, Hermansen K, Lauritzen T, Christiansen JS. Obesity does not influence the unique pharmacological properties of different biphasic insulin aspart preparations in patients with type 2 diabetes. Diabetes Obes Metab. 2010 May;12(5):414-20. doi: 10.1111/j.1463-1326.2009.01178.x. PMID 20415689
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com